CLINICAL TRIAL: NCT02348905
Title: ACTHAR Gel for Cutaneous Sarcoidosis: An Open Label Trial
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Marc A. Judson, MD, Marc A. Judson, MD, Albany Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCMAJCUT2014
Record Dates: First submitted 2014-06-20; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Sarcoidosis; Cutaneous Sarcoidosis
MeSH Terms: conditions — Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACTHAR Gel 40 units twice weekly (Experimental): ACTHAR Gel at a dose of 40 units twice weekly sub cutaneous injections between Baseline and week 12.
  Interventions: Drug: ACTHAR Gel 40 units twice weekly
- ACTHAR Gel 80 units twice weekly (Experimental): ACTHAR gel at a dose of 80 units twice weekly sub cutaneous injections between Baseline and week 12.
  Interventions: Drug: ACTHAR Gel 80 units twice weekly.

INTERVENTIONS:
Drug: ACTHAR Gel 40 units twice weekly — ACTHAR Gel (adrenocorticotropic hormone) 40 units twice weekly between Baseline and week 12.
  Arms: ACTHAR Gel 40 units twice weekly
Drug: ACTHAR Gel 80 units twice weekly. — ACTHAR Gel (adrenocorticotropic hormone) 80 units twice weekly between Baseline and week 12.
  Arms: ACTHAR Gel 80 units twice weekly

SUMMARY:
ACTHAR gel has efficacy in the treatment of cutaneous sarcoidosis

DETAILED DESCRIPTION:
Sarcoidosis is a multisystem granulomatous disease of unknown cause. Although sarcoidosis most commonly affects the lung3, it may affect any organ. Although corticosteroids are recognized as the drug of choice for sarcoidosis, ACTH is the only drug that is FDA-approved for this disorder. However, there is limited data on the efficacy of ACTH for this condition.

Presently, corticosteroids as considered the drug of choice for the treatment of cutaneous sarcoidosis. However, ACTHER GEL not only has obvious anti-inflammatory effects by resulting in corticosteroid production, but it may also activate melanocortin receptors. The melanocortin system has powerful anti-inflammatory properties that may be beneficial in the treatment of cutaneous sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have biopsy-proven sarcoidosis.
2. a) Patients with active cutaneous sarcoidosis and two active lesions on stable therapy or no therapy for at least two months AND/OR b) Patients with active cutaneous sarcoidosis and lupus pernio lesions on stable therapy or no therapy for at least two months. A maximum of 5 patients may be enrolled fulfilling criterion b) above.
3. Both lesions must have a SASI induration score of > 1 and a SASI induration + erythema score of > 2.
4. If two lesions are present, one must be > 1cm in diameter and the subject must be willing to have it biopsied. The second lesion must be at least 0.5 cm in diameter.
5. If a subject has only lupus pernio facial lesions, one needs to be at least 0.5 cm in diameter.

Exclusion Criteria:

1. Previous toxic or allergic reaction to ACTHAR gel
2. The presence of another skin condition in addition to sarcoidosis that would interfere with the assessment of the sarcoidosis skin lesions.
3. Uncontrolled hypertension.
4. Uncontrolled diabetes.
5. Active infection.
6. A medical condition that, in the opinion of the investigator would place the subject at significant risk by administering ACTHAR gel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-03; Primary Completion 2015-07 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
The change in SASI induration & erythema score. | Between week 0 and week 12.

SECONDARY OUTCOMES:
Photographic change | Between week 0 and week 12.
  Photographic change (improved, worse, no change as determined by investigators blinded to the time of the photographs)
SAT skin module | Between week 0 and week 12.
DLQI | Between week 0 and week 12.
Extent of granulomatous inflammation in the biopsy lesion | Between week 0 and week 12.
  Extent of granulomatous inflammation in the biopsy lesion (as judged by pathologists blinded to the time of the biopsy).

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Judson, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical College, Albany, New York, United States